CLINICAL TRIAL: NCT00002326
Title: A Phase I/II Study of the Safety, Tolerance, and Pharmacokinetics of Combination Zidovudine (AZT) and 9-(2-Phosphonylmethoxyethyl)Adenine (PMEA; Adefovir) Treatment in HIV-Infected Patients
Brief Title: The Safety and Effectiveness of Zidovudine Plus Adefovir in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 217B; GS-93-204
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine; Adenine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — adefovir; Zidovudine

INTERVENTIONS:
Drug: Adefovir
Drug: Zidovudine

SUMMARY:
To study the safety, tolerance, pharmacokinetics, and anti-HIV effects of combination zidovudine (AZT) and PMEA (adefovir) therapy.

DETAILED DESCRIPTION:
Patients receive AZT daily and intravenous PMEA three times weekly for 4 weeks. An MTD will be defined for this regimen.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylactic therapy with aerosolized pentamidine, oral trimethoprim/sulfamethoxazole (Bactrim, Septra) or dapsone, and fluconazole or ketoconazole IF on a stable regimen for at least 4 weeks prior to study entry.

Patients must have:

* HIV seropositivity.
* Mean CD4 count <= 500 cells/mm3.
* Been receiving AZT at 500 mg daily for at least 4 weeks prior to study entry.
* Life expectancy of at least 3 months.

NOTE:

* Kaposi's sarcoma is permitted provided patient has not received any systemic therapy for KS within the past 4 weeks. Patients with a history of another malignancy must be disease free for 6 months or more prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Inadequate venous access.
* Active, serious infections (other than HIV infection) requiring parenteral antibiotic therapy.
* Clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or clinically significant arrhythmia.
* Active malignancy other than Kaposi's sarcoma.
* Mental incapacity or illness that may affect compliance.

Concurrent Medication:

Excluded:

* ddI or ddC.
* Interferon alpha.
* Ganciclovir.
* Foscarnet.
* Diuretics.
* Investigational agents including d4T.
* Chemotherapeutic agents.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Other nephrotoxic agents.
* Immunomodulatory agents.
* Parenteral therapy for an active, serious infection (other than HIV infection).

Prior Medication:

Excluded within 2 weeks prior to study entry:

* ddI or ddC.
* Interferon alpha.
* Ganciclovir.
* Foscarnet.
* Diuretics.
* Investigational agents including d4T.
* Chemotherapeutic agents.
* Amphotericin B.
* Aminoglycoside antibiotics.
* Other nephrotoxic agents.
* Immunomodulatory agents.

Excluded within 4 weeks prior to study entry:

Systemic therapy for Kaposi's sarcoma.

Required:

* AZT at a stable dose for at least 4 weeks prior to study entry. Current use of illicit drugs (e.g., heroin or cocaine). Ingestion of substantial alcohol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (1):
- Natl Cancer Institute, Bethesda, Maryland, United States